CLINICAL TRIAL: NCT06564753
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, 13-week Study of NA-931 for Weight Management in Subjects Who Are Obese or Overweight With at Least One Weight-related Comorbid Condition
Brief Title: Phase 2 Trials of NA-931 to Study Subjects Who Are Obese With at Least One Weight-related Comorbid Condition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomed Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA-931-100
Record Dates: First submitted 2024-08-16; First posted 2024-08-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Weight Loss; Obesity; Body Weight; Body Weight Changes
Keywords: Obesity; Overweight; Weight Loss
MeSH Terms: conditions — Weight Loss; Obesity; Body Weight; Body Weight Changes; Overweight

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel arm study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo Comparator: NA-931(Placebo) (Placebo Comparator): Placebo Comparator: NA-931(Placebo) Placebo
  Interventions: Drug: Drug: Placebo daily and orally
- Experimental: NA-931 - daily orally (Dose #1) (Experimental): Experimental: NA-931 - daily orally (Dose #1) NA-931 is a peptide quadruple receptor agonist of Insulin-like Growth Hormone 1 (IGF-1), Glucagon-Like Peptide 1 (GLP-1), Glucose-dependent Insulinotropic Polypeptide (GIP), Glucagon Receptor
  Interventions: Drug: NA-931, dose 1, daily and orally
- Experimental: NA-931 - daily orally (Dose #2) (Experimental): Experimental: NA-931 - daily orally (Dose #2) NA-931 is a peptide quadruple receptor agonist of Insulin-like Growth Hormone 1 (IGF-1), Glucagon-Like Peptide 1 (GLP-1), Glucose-dependent Insulinotropic Polypeptide (GIP), Glucagon Receptor
  Interventions: Drug: NA-931, dose2, daily and orally
- Experimental: NA-931 - daily orally (Dose #3) (Experimental): Experimental: NA-931 - daily orally (Dose #3) NA-931 is a peptide quadruple receptor agonist of Insulin-like Growth Hormone 1 (IGF-1), Glucagon-Like Peptide 1 (GLP-1), Glucose-dependent Insulinotropic Polypeptide (GIP), Glucagon Receptor
  Interventions: Drug: NA-931 dose 3, daily and orally
- Experimental: NA-931 - daily orally (Dose #4) (Experimental): Experimental: NA-931 - daily orally (Dose #4) NA-931 is a peptide quadruple receptor agonist of Insulin-like Growth Hormone 1 (IGF-1), Glucagon-Like Peptide 1 (GLP-1), Glucose-dependent Insulinotropic Polypeptide (GIP), Glucagon Receptor
  Interventions: Drug: NA-931 dose 4, daily and orally

INTERVENTIONS:
Drug: Drug: Placebo daily and orally — • Placebo comparator
  Other Names: NA-931 placebo
  Arms: Placebo Comparator: NA-931(Placebo)
Drug: NA-931, dose 1, daily and orally — Drug: NA-931 dose 1, daily and orally
  • NA-931 is a peptide quadruple GLP-1, IGF-1, GIP , Glucagon quadruple agonist
  Other Names: NA-931
  Arms: Experimental: NA-931 - daily orally (Dose #1)
Drug: NA-931, dose2, daily and orally — Drug: NA-931 dose 2, daily and orally
  • NA-931 is a peptide quadruple GLP-1, IGF-1, GIP , Glucagon quadruple agonist
  Other Names: NA-931
  Arms: Experimental: NA-931 - daily orally (Dose #2)
Drug: NA-931 dose 3, daily and orally — Drug: NA-931 dose 3, daily and orally
  • NA-931 is a peptide quadruple GLP-1, IGF-1, GIP , Glucagon quadruple agonist
  Other Names: NA=931
  Arms: Experimental: NA-931 - daily orally (Dose #3)
Drug: NA-931 dose 4, daily and orally — Drug: NA-931 dose 4, daily and orally
  • NA-931 is a peptide quadruple GLP-1, IGF-1, GIP , Glucagon quadruple agonist
  Other Names: NA-931
  Arms: Experimental: NA-931 - daily orally (Dose #4)

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled, parallel arm study of NA-931 in adults who are obese (BMI ≥30 kg/m2) or who are overweight (BMI ≥27 kg/m2) with at least one weight-related co-morbid condition.

DETAILED DESCRIPTION:
This is a Phase 2, 13-week randomized, double-blind, placebo-controlled, parallel arm study that will evaluate the safety, tolerability, weight loss efficacy, pharmacodynamic effects, and pharmacokinetics of NA-931 in adults who are obese (BMI ≥30 kg/m2) or who are overweight (BMI ≥27 kg/m2) with at least one weight-related co-morbid condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age at the time of signing the informed consent
2. Body mass index (BMI) ≥30 kg/m2 or ≥27 kg/m2 with at least one weight-related co-morbid condition (treated or untreated), and BMI <50 kg/m2

Exclusion Criteria:

1. History of or current clinically significant medical or psychiatric disorder that, in the opinion of the Investigator, does not support study participation
2. Self-reported body weight change of 5% or more within 3 months of screening
3. Current or past diagnosis of diabetes mellitus (including type 1, type 2, gestational)
4. Current or past diagnosis of chronic pancreatitis
5. Calcitonin ≥20 ng/L measured by central laboratory at screening (individuals with elevated calcitonin at initial screening may be re-screened)
6. Any Glucagon-Like Peptide 1 (GLP-1) receptor agonist or GLP-1/ Glucose-dependent Insulinotropic Polypeptide (GIP) dual agonist within 6 months of Screening
7. Any prescription or over-the-counter medications intended for weight loss within 6 months of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Percent (relative) change from baseline to Week 13 in body weight | 13 weeks
  To measure the efficacy of NA-931 for weight loss in adult subjects who are obese, or overweight with at least one weight-related comorbid condition

SECONDARY OUTCOMES:
Proportion of Subjects losing ≥5% and ≥10% of baseline weight at Week 13 | 13 weeks
  To measure the efficacy of NA-931 for weight loss in adult subjects who are obese, or overweight with at least one weight-related comorbid condition
Incidence of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse event (TESAEs), adverse events of special interest (AESI) | 13 weeks
  To evaluate the safety and tolerability including treatment-emergent adverse events (TEAEs), TESAEs, AESI of NA-931 for weight loss in adult subjects who are obese, or overweight with at least one weight-related comorbid condition

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Tran, PhD, Principal Investigator — Biomed Industries, Inc.
Locations (5):
- Australia (5):
  - Biomed Investigational Site, Camperdown, New South Wales
  - Biomed Investigational Site, Merewether, New South Wales
  - Biomed Investigational Site, St Leonards, New South Wales
  - Biomed Investigational Site, Heidelberg Heights, Victoria
  - Biomed Investigational Site, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
The investigators plan to share individual participant data (IPD) available to other researchers.